CLINICAL TRIAL: NCT01667263
Title: The Combination of Oral All-trans Retinoic Acid and Danazol vs Danazol as Second-line Treatment in Adult Immune Thrombocytopenia: a Multicenter, Randomized, Open-label Trial
Brief Title: The Combination of ATRA and Danazol as Second-line Treatment in Adult Immune Thrombocytopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other); Beijing Hospital (Other Government); Qilu Hospital of Shandong University (Other); Navy General Hospital, Beijing (Other); Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Xiao-hui Zhang, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1132-6877; Z111107058811024 (Other Grant/Funding Number: Capital Clinical characteristic application foundation)
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-04

CONDITIONS: Autoimmune Thrombocytopenia
Keywords: All-trans retinoic acid; primary immune thrombocytopenia; corticosteroid-resistant; refractory; danazol
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Tretinoin; Danazol; deanol aceglutamate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- All-trans retinoic acid ＆Danazol (Experimental): Danazol 400mg po and ATRA 10mg bid po
  Interventions: Drug: All-trans retinoic acid; Drug: Danazol
- Danazol (Active Comparator): Danazol 400mg po
  Interventions: Drug: Danazol

INTERVENTIONS:
Drug: All-trans retinoic acid
  Other Names: Retinoid acid
  Arms: All-trans retinoic acid ＆Danazol
Drug: Danazol
  Other Names: Danocrine; Cleregil; Danol

SUMMARY:
Randomized, open-label, multicentre study to compare the efficacy and safety of ATRA plus danazol with danazol monotherapy in patients with corticosteroid-resistant/relapsed ITP.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is a severe bleeding disorder. Approximately 2/3 of patients achieve remission from first-line therapies. However, the underlying mechanism of corticosteroid-resistant or relapsed ITP is not well understood; thus, treatment remains a great challenge. All-trans retinoic acid (ATRA) has an immunomodulatory effect on haematopoiesis, making it a possible treatment option.

A multicentre prospective study was performed in non-splenectomized ITP patients who were either resistant to a standard dose of corticosteroids or had relapsed. Patients were randomized to ATRA+danazol and danazol monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study, in order to compare the efficacy and safety of ATRA plus danazol with danazol monotherapy in patients with corticosteroid-resistant/relapsed ITP.

ELIGIBILITY:
Inclusion Criteria:

* Primary immune thrombocytopenia (ITP) confirmed by excluding other supervened causes of thrombocytopenia;
* Platelet count of less than 30×109/L at enrolment
* Patients who did not achieve a sustained response to treatment with full-dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid-tapering or after its discontinuation.
* 18 years older.

Exclusion Criteria:

* Secondary immune thrombocytopenia (e.g., patients with HIV, HCV, Helicobacter pylori infection or patients with systemic lupus erythematosus)
* congestive heart failure
* severe arrhythmia
* nursing or pregnant women
* aspartate aminotransferase and alanine transaminase levels ≥ 3× the upper limit of the normal threshold criteria
* creatinine or serum bilirubin levels each 1•5 times or more than the normal range
* active or previous malignancy
* Unable to do blood routine test for the sake of time, distance, economic issues or other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
the sustained platelet response at the 12-month follow-up | From the start of study treatment (Day 1) up to the end of Month 12
  The number of participants (responders) with platelet count >=30x10^9/L and at least a 2-fold increase in the baseline count (PR) or a platelet count >=100x10^9/L (CR) and the absence of bleeding, without rescue medication at 12-month follow-up.

SECONDARY OUTCOMES:
overall response | From the start of study treatment (Day 1) up to the end of Month 12
  The number of participants with platelet count >=30×10^9/L at least once and at least a doubling of the baseline platelet count without the administration of any other platelet increasing therapy
primary response rate at 4 weeks | From the start of study treatment (Day 1) up to week 4 of treatment
  The number of participants with platelet count >=30×10^9/L and at least a doubling of the baseline platelet count without the administration of any other platelet increasing therapy at week 4 of treatment
primary response rate at 8 weeks | From the start of study treatment (Day 1) up to week 8 of treatment
  The number of participants with platelet count >=30×10^9/L and at least a doubling of the baseline platelet count without the administration of any other platelet increasing therapy at week 8 of treatment
time to response | From the start of study treatment (Day 1) up to the end of month 12
  Time to response was defined as the time from starting treatment to the time to achieve the response.
duration of response | From the start of study treatment (Day 1) up to the end of month 12
  Duration of response was measured from the achievement of response to the loss of response.
reduction in bleeding symptoms | From the start of study treatment (Day 1) up to the end of month 12
  Changes of bleeding after treatment. Bleeding was defined in accordance with the WHO bleeding scale (0, no bleeding; 1, petechiae; 2, mild blood loss; 3, gross blood loss; and 4, debilitating blood loss).
safety | From the start of study treatment (Day 1) up to the end of follow-up
  All patients were assessed for safety every week during the first 8 weeks of treatment, and at 2-week intervals thereafter. Adverse events were scaled according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, Professor, Principal Investigator — Peking University People's Hospital, Peking University Insititute of Hematology
Locations (5):
- China (5):
  - Beijing Hospital, Ministry of Health, Beijing, Beijing Municipality
  - Peking University People's Hospital, Peking University Insititute of Hematology, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - PLA Navy General Hospital, Beijing, Beijing Municipality
  - Qilu Hospital, Shandong University, Jinan, Shandong

REFERENCES:
- [Background] Zhang X, Fu H, Xu L, Liu D, Wang J, Liu K, Huang X. Prolonged thrombocytopenia following allogeneic hematopoietic stem cell transplantation and its association with a reduction in ploidy and an immaturation of megakaryocytes. Biol Blood Marrow Transplant. 2011 Feb;17(2):274-80. doi: 10.1016/j.bbmt.2010.09.007. Epub 2010 Sep 18. PMID 20854919
- [Background] Nozaki Y, Tamaki C, Yamagata T, Sugiyama M, Ikoma S, Kinoshita K, Funauchi M. All-trans-retinoic acid suppresses interferon-gamma and tumor necrosis factor-alpha; a possible therapeutic agent for rheumatoid arthritis. Rheumatol Int. 2006 Jul;26(9):810-7. doi: 10.1007/s00296-005-0076-1. Epub 2005 Nov 15. PMID 16292516
- [Background] Sakakura M, Wada H, Tawara I, Nobori T, Sugiyama T, Sagawa N, Shiku H. Reduced Cd4+Cd25+ T cells in patients with idiopathic thrombocytopenic purpura. Thromb Res. 2007;120(2):187-93. doi: 10.1016/j.thromres.2006.09.008. Epub 2006 Oct 24. PMID 17067661
- [Background] Wang ZY, Chen Z. Acute promyelocytic leukemia: from highly fatal to highly curable. Blood. 2008 Mar 1;111(5):2505-15. doi: 10.1182/blood-2007-07-102798. PMID 18299451
- [Background] Wing K, Larsson P, Sandstrom K, Lundin SB, Suri-Payer E, Rudin A. CD4+ CD25+ FOXP3+ regulatory T cells from human thymus and cord blood suppress antigen-specific T cell responses. Immunology. 2005 Aug;115(4):516-25. doi: 10.1111/j.1365-2567.2005.02186.x. PMID 16011520
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Background] LIU Wen-bin, WANG Zhao-yue, CAO Li-juan, ZHAO Xiao-juan, ZHU Ming-qing, BAI Xia, RUAN Chang-geng.Therapeutic Effect and Mechanism of All-trans-retinoic Acid Treatment in Refractory Idiopathic Thrombocytopenic Purpura.Suzhou University Journal of Medical Science.2009;3 476-479.
- [Derived] Feng FE, Feng R, Wang M, Zhang JM, Jiang H, Jiang Q, Lu J, Liu H, Peng J, Hou M, Shen JL, Wang JW, Xu LP, Liu KY, Huang XJ, Zhang XH. Oral all-trans retinoic acid plus danazol versus danazol as second-line treatment in adults with primary immune thrombocytopenia: a multicentre, randomised, open-label, phase 2 trial. Lancet Haematol. 2017 Oct;4(10):e487-e496. doi: 10.1016/S2352-3026(17)30170-9. Epub 2017 Sep 13. PMID 28917657